CLINICAL TRIAL: NCT03664440
Title: Efficacy of Rilpivirine-based Regimens as Switch Therapy From Nevirapine-based Regimens in HIV-infected Patients With Complete Virological Suppression: A Randomized Controlled Trial
Brief Title: Efficacy of Rilpivirine-based Regimens as Switch Therapy From Nevirapine-based Regimens in HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-59-04
Record Dates: First submitted 2018-08-16; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Efficacy of Rilpivirine-based Regimens as Switch Therapy
Keywords: rilpivirine switch therapy
MeSH Terms: interventions — Nevirapine; Rilpivirine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuation arm (Placebo Comparator): patients who currently received TDF/3TC/NVP (group A) or TDF/FTC/NVP (group B) were block 4 randomly assigned (1:1) by computer-generated random numbers, to continue their current regimen of NVP 200 mg twice daily plus TDF/3TC (group A1) and plus TDF/FTC (groupB1)
  Interventions: Drug: Nevirapine
- switch arm (Active Comparator): patients who currently received TDF/3TC/NVP (group A) or TDF/FTC/NVP (group B) were block 4 randomly assigned (1:1) by computer-generated random numbers to switch from NVP to RPV 25 mg once-daily plus TDF/3TC (group A2) and plus TDF/FTC (groupB2)
  Interventions: Drug: Rilpivirine

INTERVENTIONS:
Drug: Nevirapine — Patients were randomized 1:1 to continuation arm (NVP-based regimens). Tenofovir disoproxil fumarate (TDF) plus lamivudine (3TC) or emtricitabine (FTC) remained as the backbone of the regimens.
  Arms: continuation arm
Drug: Rilpivirine — Patients were randomized 1:1 to switch arm (NVP-based regimens were switched to RPV-based regimens). Tenofovir disoproxil fumarate (TDF) plus lamivudine (3TC) or emtricitabine (FTC) remained as the backbone of the regimens.
  Arms: switch arm

SUMMARY:
Background: Nevirapine (NVP)-based antiretroviral therapy (ART) remains to be used in HIV-infected patients in resource limited countries despite its compliance and adverse effect concerns. Rilpivirine (RPV), a newer non-nucleoside reverse transcriptase inhibitor, could be used as an alternative to NVP in virologically suppressed patients. However, there has been limited experience with switching from NVP-based to RPV-based regimens. The investigators aimed to study efficacy and adverse events after ART switching from NVP-based to RPV-based regimens.

Methods: A randomized controlled non-inferiority trial was conducted in HIV-infected patients who received NVP-based regimens and had undetectable plasma HIV RNA for more than 6 months. Patients were randomized 1:1 to continuation arm (NVP-based regimens were continued) or switch arm (NVP-based regimens were switched to RPV-based regimens). Tenofovir disoproxil fumarate (TDF) plus lamivudine (3TC) or emtricitabine (FTC) remained as the backbone of the regimens. Primary endpoint was HIV RNA <40 copies/mL at 48 weeks, with a non-inferiority margin of 12%. Changes of CD4 cell counts and lipid profiles from baseline were analyzed.

DETAILED DESCRIPTION:
A single-center randomized controlled, non-inferiority trial to study 48-week treatment outcomes of RPV as a switch therapy was conducted at Ramathibodi Hospital, a tertiary care health center in Thailand from December 2016 to October 2017 Eligible patients who currently received TDF/3TC/NVP (group A) or TDF/FTC/NVP (group B) were block 4 randomly assigned (1:1) by computer-generated random numbers, to continue their current regimen of NVP 200 mg twice daily plus TDF/3TC (group A1) and plus TDF/FTC (groupB1), or to switch from NVP to RPV 25 mg once-daily plus TDF/3TC (group A2) and plus TDF/FTC (groupB2). Patients were advised to take RPV with a meal. Patients were scheduled trial visits at baseline, week 12, 24, 36 and week 48. The laboratory assessment was performed at baseline week 24 and week 48.

ELIGIBILITY:
Inclusion Criteria:

* Recent plasma HIV-1 RNA viral load within 6 months of the screening that was less than 40 copies/mL, and a CD4 cell count that was more than 200 cells/mm3
* Patient who treated with TDF/FTC/NVP or TDF/3TC/NVP for at least 6 month

Exclusion Criteria:

* patients with a history of HIV drug resistance, patients who used other drugs or drugs which interact with RPV (proton pump inhibitors, histamine H2-receptor antagonists, rifampin, antiepileptic drugs), female patients during pregnancy or breastfeeding, patients whose estimated glomerular filtration rate (eGFR)was <60 mL/min/1.73m2 [by The Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) (12)], and patients diagnosed with depressive or psychiatric disorders.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
HIV RNA viral load | week 48
  HIV-1 RNA viral load was performed at 48 by using Amplicor HIV-1 Monitor Test version 1.5 (Roche, Basel, Switzerland)

SECONDARY OUTCOMES:
CD4 cell count | week 48
  blood for CD4 cell count was performed at week 48
CD4 percentage | week 48
  blood for CD4 percentage was performed at week 48
Change of total cholesterol | baseline and week 48
  Change from baseline of total cholesterol was performed at week 48
Change of high-density lipoprotein cholesterol level (HDL-c) | baseline and week 48
  Change from baseline of high-density lipoprotein cholesterol level (HDL-c) was performed at week 48
Change of low-density lipoprotein cholesterol level (LDL-c) | baseline and week 48
  Change from baseline of low-density lipoprotein cholesterol level (LDL-c) was performed at week 48
Change of triglyceride | baseline and week 48
  Change from baseline of triglyceride was performed at week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Hagins D, Orkin C, Daar ES, Mills A, Brinson C, DeJesus E, Post FA, Morales-Ramirez J, Thompson M, Osiyemi O, Rashbaum B, Stellbrink HJ, Martorell C, Liu H, Liu YP, Porter D, Collins SE, SenGupta D, Das M. Switching to coformulated rilpivirine (RPV), emtricitabine (FTC) and tenofovir alafenamide from either RPV, FTC and tenofovir disoproxil fumarate (TDF) or efavirenz, FTC and TDF: 96-week results from two randomized clinical trials. HIV Med. 2018 Nov;19(10):724-733. doi: 10.1111/hiv.12664. Epub 2018 Aug 12. PMID 30101539
- [Background] Taramasso L, Tatarelli P, Ricci E, Madeddu G, Menzaghi B, Squillace N, De Socio GV, Martinelli C, Gulminetti R, Maggi P, Orofino G, Vichi F, Di Biagio A, Bonfanti P; CISAI Study Group. Improvement of lipid profile after switching from efavirenz or ritonavir-boosted protease inhibitors to rilpivirine or once-daily integrase inhibitors: results from a large observational cohort study (SCOLTA). BMC Infect Dis. 2018 Jul 31;18(1):357. doi: 10.1186/s12879-018-3268-5. PMID 30064371